CLINICAL TRIAL: NCT00183989
Title: A Pilot Phase II Trial of Combination Therapy With Fludarabine, Mitoxantrone and Rituximab in Mantle Cell Lymphoma
Brief Title: Combination Therapy With Fludarabine, Mitoxantrone and Rituximab in Mantle Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13NHL-99-2
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — fludarabine; Mitoxantrone; Rituximab

INTERVENTIONS:
Drug: Fludarabine, Mitoxantrone and Rituximab

SUMMARY:
This study is being done in order to determine the effectiveness of the combination of fludarabine, mitoxantrone, and rituximab in patients with mantle cell lymphoma. All three drugs,fludarabine, mitoxantrone, and rituximab have been approved by the U.S. Food and Drug Administration (FDA)for the treatment of certain types of lymphoma. Rituximab is a drug (called a monoclonal antibody) which has anti-tumor activity on certain types of lymphoma. The combination of chemotherapy (fludarabine and mitoxantrone) with rituximab has not yet been investigated in patients with mantle cell lymphoma and therefore the combination in investigational.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of Non-Hodgkin's Lymphoma of the mantle cell sub-type lymphoma only, as determined by morphologic assessment and consistent immunophemotypic markers
* Newly diagnosed and patients who have received prior treatment are eligible
* Measurable or evaluable disease
* Karnofsky performance status greater or equal to 50%
* Men and women, age greater or equal to 18 years old
* AGC greater or equal to 1.0; platelets greater or equal to 75,000; Hemoglobin greater or equal to 8.0 (unless because of lymphomatous infiltration of the marrow)
* Creatinine less than 2.0; bilirubin less than 2.0; SGOT less than 3 times upper limit of normal (unless elevations are due to lymphomatous involvement)
* Women of child bearing potential must have negative pregnancy test within 14 days of study entry.
* Signed informed consent

Exclusion Criteria:

* History of congestive heart failure or significant cardiac disease
* Prior exposure to either fludarabine or mitoxantrone. Prior exposure to rituximab allowed
* Active infection
* HIV seropositive
* Pregnant or lactating females
* Second active malignancy, other than squamous cell skin cancer,in-situ cervical cancer, or history of other cancer diagnosed within the preceding 5 years
* Presence of psychological or emotional disorders which would make valid informed consent impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2000-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra M. Levine, MD, Principal Investigator — University of Southern California
Locations (1):
- Norris Comprehensive Cancer Center, Los Angeles, California, United States